CLINICAL TRIAL: NCT06806995
Title: A Single-center, Open-label, Study Evaluating Safety and Pharmacokinetics of Single Doses of Zidebactam-Cefepime and Metronidazole Alone or in Combination Utilizing a 3-Period, Crossover Study Design
Brief Title: A Single-center, Open-label, Study Evaluating Safety and Pharmacokinetics of Single Doses of Zidebactam-Cefepime and Metronidazole Alone or in Combination.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wockhardt (Industry)
Collaborators: Eric Solutions LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: W-5222-106
Record Dates: First submitted 2025-01-15; First posted 2025-02-04 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-01

CONDITIONS: PHA1A
MeSH Terms: interventions — cefepime-zidebactam; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zidebactam Cefepime (Experimental): Zidebactam Cefepime 3gm Vial
  Interventions: Drug: Zidebactam-Cefepime; Drug: Metronidazole; Drug: FEP-ZID

INTERVENTIONS:
Drug: Zidebactam-Cefepime — (1) ZID-FEP 3g IV (ZID 1 g plus FEP 2 g) administered over 1 hour (h)
Drug: Metronidazole — (2) metronidazole 0.5 g IV alone administered over 1 h
Drug: FEP-ZID — (3) metronidazole 0.5 g IV over 1 h, followed by ZID-FEP 3g IV over 1 h over 3 treatment periods separated by a 48 h washout period.

SUMMARY:
This is a Phase I, Single-Center, Open-Label study evaluating the safety and pharmacokinetics of single doses of ZID-FEP and metronidazole alone or in combination utilizing a 3-period, crossover study design. Thirty eligible male and female healthy adult subjects will participate in the study and receive single doses of (1) ZID-FEP 3g IV (ZID 1 g plus FEP 2 g) administered over 1 hour (h); (2) metronidazole 0.5 g IV alone administered over 1 h; and (3) metronidazole 0.5 g IV over 1 h, followed by ZID-FEP 3g IV over 1 h over 3 treatment periods separated by a 48 h washout period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 45 years of age (inclusive)
2. Body mass index of 18 to 31 kg/m2 (inclusive).
3. Subjects voluntarily consented to participate in this study and who have signed and dated the informed consent form.
4. No major pathology/surgery in the 6 months prior to screening Agrees to use effective methods of contraception
5. Resting supine blood pressure of 90 to 139 (systolic)/50 to 89 (diastolic) mmHg and a resting pulse rate of 40 to 100 beats per minute.
6. Calculated creatinine clearance ≥90 mL/min (Cockcroft-Gault method).
7. Computerized 12-lead ECG recording without signs of clinically significant pathology and showing no clinically significant deviation as judged by the Principal Investigator. The QT interval corrected for heart rate using Fridericia's formula must be ≤450 ms for males and be ≤460 ms for females.
8. Males must agree not to donate sperm and if engaging in sexual intercourse with a female partner who could become pregnant, must agree to use a condom and highly effective method of contraception (see Section 6.6) until 90 days after the last administration of study drug.
9. Females should not be pregnant or breastfeeding (to be confirmed by a urine pregnancy test at screening with confirmation by a serum pregnancy test at admission) or should be of non-childbearing potential at screening.
10. Females must be either postmenopausal for at least 1 year, surgically sterile (bilateral oophorectomy or hysterectomy), or practicing one of the acceptable methods of birth control, as defined in inclusion criteria #7, for 3 weeks prior to study drug administration, during the study, and for 90 days after the last administration of study drug.
11. All values of hematology, serum chemistry, coagulation, and urinalysis showing no clinically significant deviations from the normal range as judged by the Principal Investigator.

Exclusion Criteria:

1. Participation in another investigational drug or device study or treated with a study drug within 30 days or 5 half-lives, whichever is longer, before receiving any study drug in this study.
2. History/evidence of clinically relevant pathology related to the cardiovascular system, central nervous system, respiratory tract, gastrointestinal tract, endocrinology, immunology, hematology or any other systemic disorder/major surgeries, that in the opinion of the Principal Investigator would confound the subject's participation and follow-up in the study.
3. History of clinically significant food or drug allergy, including known hypersensitivity to cefepime or metronidazole or any other related drugs.
4. History of Clostridium difficile induced diarrhea or infection within 1 year before screening.
5. Prior exposure to zidebactam.
6. Consumed more than 28 units of alcohol per week at any time in the 6 months before study drug administration (1 unit of alcohol is equivalent to 8 ounces of beer, 4 ounces of wine, or 1 ounce of spirits) or history of active alcoholism and/or drug/chemical abuse within the last 3 to 5 years.
7. A positive screen result for drugs of abuse/alcohol at admission to the study center at Check-in.
8. Use of prescription medications (with the exception of oral contraceptives, all forms of hormonal contraceptives, and hormone replacement therapy) including nonsteroidal anti-inflammatory drugs or sucralfate or herbal preparations within 14 days or 5 half-lives (whichever is longer) before study drug administration, or use of over-the-counter medication, acetaminophen (>500 mg/day), vitamins, or supplements (including fish liver oils) within 7 days before the first administration of study drug. Acetaminophen ≤500 mg/day is allowable 3 days before enrollment in the study (Day 1). Should the subject have taken any other medications the Investigator will discuss enrolling the subject with the medical monitor on a case-by-case basis.
9. Positive serology test for hepatitis B surface antigen, hepatitis C virus or human immunodeficiency virus I/II at screening.
10. Any strenuous activity within 96 hours (4 days) prior to enrollment in the study. Strenuous is defined as any hard labor or exercise outside of a subject's usual behavior.
11. Unable or unwilling to stay in the study center for the required duration as per the protocol or consume the standard meal provided by the study center.
12. History of blood donation of more than 500 mL in the last 2 months prior to screening.
13. Consumption of methylxanthine-containing food or beverages (such as coffee, tea, cola, chocolate, 'power drinks'), grapefruit or grapefruit juice, or Seville oranges or products containing Seville oranges for 48 hours prior to enrollment in the study and while resident at the study center.
14. Current use or has used tobacco- or nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, etc.) 30 days prior to study drug administration. A cotinine test (with a cut-off of 200 mg) will be performed at screening and at Check-In (Day -1).
15. Subject has a history of difficulty in providing blood samples or has poor veins which may cause difficulty in obtaining blood samples during the study.
16. History of bleeding disorders.
17. Unable or unwilling to follow study instruction or restrictions or a history of the same.
18. Any other medical, psychological, or social condition which, in the opinion of the Principal Investigator would prevent the subject from fully participating in the study, would represent a concern for study compliance, or would constitute a safety concern for the subject.
19. Any person who is an employee of the Principal Investigator or study center with direct involvement in this proposed study or any other study under the direction of the Principal Investigator or the study center or who is directly involved in the planning and/or conduct of the study, as well as relatives of the employee, the Investigators, or the Sponsor.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
To assess Plasma Pharmacokinetics Parameters | Day 1, 4, 7
  Maximum concentration (Cmax)
To assess Plasma Pharmacokinetics Parameters | Day 1, 4, 7
  Area under the concentration time curve up to infinity (AUC0-inf) for each analyte

SECONDARY OUTCOMES:
To Assess Plasma Pharmacokinetics Parameters Area Under Concentration | Day 1, 4, 7
  Area Under Concentration Time curve up to last measurable time point (AUClast)
To Assess Plasma Pharmacokinetics Parameters Time to reach maximum concentration | Day 1, 4, 7
  Time to reach maximum concentration (Tmax)
To Assess Plasma Pharmacokinetics Parameters Terminal elimination half-life | Day 1, 4, 7
  Terminal elimination half-life (T½)
To Assess Plasma Pharmacokinetics Parameters Plasma Clearance | Day 1, 4, 7
  Plasma Clearance (CL)
To Assess Plasma Pharmacokinetics Parameters Volume of Distribution | Day 1, 4, 7
  Volume of Distribution (Vz)

OTHER OUTCOMES:
Protein Binding | Day 1, 4, 7
  Protein binding for cefepime and zidebactam when ZID-FEP is administered alone
Measurement of Plasma PK Parameters | Day 1, 4, 7
  Serial blood samples will be collected from all subjects for determination of drug concentration-time profiles and PK parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Pharma CR, LLC, Miami, Florida, United States